CLINICAL TRIAL: NCT03291587
Title: Implementation Of Smoking Cessation Services Within NCI NCORP Community Sites With Organized Lung Cancer Screening Programs
Brief Title: Implementation of Smoking Cessation Within NCI Community Oncology Research Program (NCORP) Sites
Acronym: OaSiS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00040071; 1R01CA207158-01 (NIH); REBAWF-20817CD (Other: NCI); NCI-2017-01669 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Smoking Cessation
Keywords: lung cancer; cancer screening; tobacco use
MeSH Terms: conditions — Smoking Cessation; Lung Neoplasms; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Training of Lung Cancer Screening Personnel on implementation of the United States Public Health Service (US PHS) Guidelines for Smoking Cessation and Performance Coaching during Implementation Phase of the Study
  Data collection from Patients: demographics, health status, smoking history, quitting behavior, perceptions of lung cancer risk and worry, impact of screening on tobacco use behavior, and exposure to the intervention. (baseline, <14 days, 3 months, and 6 months)
  Interventions: Other: Personnel Training and Coaching Calls
- Usual Care (No Intervention): No training or performance coaching calls on personnel, just usual clinic practice.
  Data collection from Patients: demographics, health status, smoking history, quitting behavior, perceptions of lung cancer risk and worry, impact of screening on tobacco use behavior, and exposure to the intervention. (baseline, <14 days, 3 months, and 6 months)

INTERVENTIONS:
Other: Personnel Training and Coaching Calls — Training of Lung Cancer Screening Personnel on implementation of the US PHS Guidelines for Smoking Cessation and Performance Coaching during Implementation Phase of the Study
  Each site will have a coaching team: two members of our research team including an expert in tobacco cessation and an expert in lung cancer screening. Active coaching includes six, 1-1 ½ hour video exchanges among program sites and coaching teams, once every 4-6 weeks over an 8-month implementation phase. One week prior to the call, each site will be prompted with an email to inform the coaching team of any challenges associated with implementation.
  Arms: Intervention

SUMMARY:
Evaluate a multi-faceted training program to improve short-term smoking cessation rates (<14 days post-visit) and short (3 months) and sustained abstinence (6 months) among 1,114 enrolled smokers who present for low-dose computed tomography (LDCT) lung cancer screening in 26 community-based practices.

DETAILED DESCRIPTION:
We utilize an effectiveness-implementation hybrid design, employing a cluster, randomized control trial of community-based NCORP sites to study the effectiveness of a multi-faceted intervention to improve smoking cessation among lung cancer screening patients, as well as dissemination and implementation (D&I) science to optimize and accelerate translation of findings into clinical practice. We will: (1) Evaluate a multi-faceted training program to improve short-term smoking cessation rates (1-week post-visit) and sustained abstinence (6 months) among 1,114 enrolled smokers (557 in each trial arm) who present for LDCT lung cancer screening in community-based lung cancer screening practices; (2) Characterize the adoption and adaptation of the evidence-based tobacco cessation strategies in 26 community-based LDCT lung cancer screening programs; and (3) Develop and evaluate an implementation toolkit for integrating evidence-based tobacco cessation strategies in community-based LDCT lung cancer screening programs. Qualitative data will be collected from key informants at participating screening programs during and after intervention implementation. Quantitative survey data (baseline, <14 days, 3 months, and 6 months) and saliva specimens (6 months only) will be collected from smoking patients receiving screening within these programs.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to have NCORP research personnel serve as the study liaison and another person to serve as the cessation program champion.
* Agrees to participate in all aspects of the intervention, randomization, and evaluation.
* Agrees to participate in a confidential 1-on-1 semi-structured interview with the research team.
* Agrees to have the interview taped, transcribed and qualitatively analyzed.
* Age ≥18 years
* Potential participants will be screened using the following question: "Do you smoke cigarettes every day, some days, or not at all?" (BRFSS). A current smoker is anyone responds "every day" or "some days".

Exclusion Criteria:

* Current use (previous 30 days) of a tobacco dependence treatment including bupropion, varenicline, and nicotine replacement
* Individuals who use e-cigarettes and who are not smoking cigarettes. Dual users (those who use both e-cigarettes and cigarettes) will still be included in the trial.
* The presence of a physical or cognitive impairment that would prevent a person from engaging in survey research (such as blindness, deafness, or dementia).
* Individual has already completed the intended LDCT lung cancer screening for this study.
* Non-English speaking participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1094 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Foley, PhD, Study Chair — Wake Forest University Health Sciences
Locations (49):
- United States (49):
  - Helen F Graham Cancer Center, Newark, Delaware
  - Augusta University Medical Center, Augusta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ridgeview Medical Center, Waconia, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest (WF) NCORP Research Base (RB) is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI National Clinical Trials Network (NCTN)/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials (https://nctn-data-archive.nci.nih.gov/). This will become the primary means for sharing raw data and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide.
Time Frame: see NIH policy
Access Criteria: request using uniform resource locator (URL) below
URL: https://nctn-data-archive.nci.nih.gov/

REFERENCES:
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Taylor DH Jr, Hasselblad V, Henley SJ, Thun MJ, Sloan FA. Benefits of smoking cessation for longevity. Am J Public Health. 2002 Jun;92(6):990-6. doi: 10.2105/ajph.92.6.990. PMID 12036794
- [Background] Hermanson B, Omenn GS, Kronmal RA, Gersh BJ. Beneficial six-year outcome of smoking cessation in older men and women with coronary artery disease. Results from the CASS registry. N Engl J Med. 1988 Nov 24;319(21):1365-9. doi: 10.1056/NEJM198811243192101. PMID 3185646
- [Background] Gellert C, Schottker B, Brenner H. Smoking and all-cause mortality in older people: systematic review and meta-analysis. Arch Intern Med. 2012 Jun 11;172(11):837-44. doi: 10.1001/archinternmed.2012.1397. PMID 22688992
- [Background] Parsons A, Daley A, Begh R, Aveyard P. Influence of smoking cessation after diagnosis of early stage lung cancer on prognosis: systematic review of observational studies with meta-analysis. BMJ. 2010 Jan 21;340:b5569. doi: 10.1136/bmj.b5569. PMID 20093278
- [Background] Black WC, Gareen IF, Soneji SS, Sicks JD, Keeler EB, Aberle DR, Naeim A, Church TR, Silvestri GA, Gorelick J, Gatsonis C; National Lung Screening Trial Research Team. Cost-effectiveness of CT screening in the National Lung Screening Trial. N Engl J Med. 2014 Nov 6;371(19):1793-802. doi: 10.1056/NEJMoa1312547. PMID 25372087
- [Background] McMahon PM, Kong CY, Bouzan C, Weinstein MC, Cipriano LE, Tramontano AC, Johnson BE, Weeks JC, Gazelle GS. Cost-effectiveness of computed tomography screening for lung cancer in the United States. J Thorac Oncol. 2011 Nov;6(11):1841-8. doi: 10.1097/JTO.0b013e31822e59b3. PMID 21892105
- [Background] Zeliadt SB, Heffner JL, Sayre G, Klein DE, Simons C, Williams J, Reinke LF, Au DH. Attitudes and Perceptions About Smoking Cessation in the Context of Lung Cancer Screening. JAMA Intern Med. 2015 Sep;175(9):1530-7. doi: 10.1001/jamainternmed.2015.3558. PMID 26214612
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for lung cancer: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2014 Mar 4;160(5):330-8. doi: 10.7326/M13-2771. PMID 24378917
- [Background] Ostroff JS, Copeland A, Borderud SP, Li Y, Shelley DR, Henschke CI. Readiness of Lung Cancer Screening Sites to Deliver Smoking Cessation Treatment: Current Practices, Organizational Priority, and Perceived Barriers. Nicotine Tob Res. 2016 May;18(5):1067-75. doi: 10.1093/ntr/ntv177. Epub 2015 Sep 7. PMID 26346948
- [Background] Clinical Practice Guideline Treating Tobacco Use and Dependence 2008 Update Panel, Liaisons, and Staff. A clinical practice guideline for treating tobacco use and dependence: 2008 update. A U.S. Public Health Service report. Am J Prev Med. 2008 Aug;35(2):158-76. doi: 10.1016/j.amepre.2008.04.009. PMID 18617085
- [Background] Tong EK, Strouse R, Hall J, Kovac M, Schroeder SA. National survey of U.S. health professionals' smoking prevalence, cessation practices, and beliefs. Nicotine Tob Res. 2010 Jul;12(7):724-33. doi: 10.1093/ntr/ntq071. Epub 2010 May 27. PMID 20507899
- [Background] Okuyemi KS, Reitzel LR, Fagan P. Interventions to Reduce Tobacco-Related Health Disparities. Nicotine Tob Res. 2015 Aug;17(8):887-91. doi: 10.1093/ntr/ntv096. No abstract available. PMID 26180213
- [Background] Foley KL, Pockey JR, Helme DW, Song EY, Stewart K, Jones C, Spangler JG, Sutfin EL. Integrating evidence-based tobacco cessation interventions in free medical clinics: opportunities and challenges. Health Promot Pract. 2012 Sep;13(5):687-95. doi: 10.1177/1524839911433465. Epub 2012 Mar 30. PMID 22467664
- [Background] Pockey JR, Song EY, Sutfin EL, Spangler JG, Jones C, Helme DW, Foley KL. The need for tobacco cessation in a free clinic population. Addict Behav. 2012 Dec;37(12):1299-302. doi: 10.1016/j.addbeh.2012.03.032. Epub 2012 Jul 4. PMID 22958861
- [Background] Error in Text and Table. Primary Care Provider-Delivered Smoking Cessation Interventions and Smoking Cessation Among Participants in the National Lung Screening Trial. JAMA Intern Med. 2015 Sep;175(9):1587-8. doi: 10.1001/jamainternmed.2015.4006. No abstract available. PMID 26348525
- [Background] Fiore MC, Goplerud E, Schroeder SA. The Joint Commission's new tobacco-cessation measures--will hospitals do the right thing? N Engl J Med. 2012 Mar 29;366(13):1172-4. doi: 10.1056/NEJMp1115176. Epub 2012 Mar 14. No abstract available. PMID 22417200
- [Background] G.A. Colditz. The promise and challenges of dissemination and implementation research. In: Dissemination and Implementation Research in Health. New York: Oxford University Press; 2012.
- [Background] Balas EA, Boren SA. Managing Clinical Knowledge for Health Care Improvement. Yearb Med Inform. 2000;(1):65-70. No abstract available. PMID 27699347
- [Background] Brownson RC, Jones E. Bridging the gap: translating research into policy and practice. Prev Med. 2009 Oct;49(4):313-5. doi: 10.1016/j.ypmed.2009.06.008. Epub 2009 Jun 22. PMID 19555708
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Goulart BH, Ramsey SD. Moving beyond the national lung screening trial: discussing strategies for implementation of lung cancer screening programs. Oncologist. 2013;18(8):941-6. doi: 10.1634/theoncologist.2013-0007. Epub 2013 Jul 19. PMID 23873718
- [Background] Marcus PM. Lung cancer screening with low dose computed tomography (LDCT): looking back and moving forward. Ann Transl Med. 2015 May;3(Suppl 1):S41. doi: 10.3978/j.issn.2305-5839.2015.03.36. No abstract available. PMID 26046089
- [Background] Kent EE, Mitchell SA, Castro KM, DeWalt DA, Kaluzny AD, Hautala JA, Grad O, Ballard RM, McCaskill-Stevens WJ, Kramer BS, Clauser SB. Cancer Care Delivery Research: Building the Evidence Base to Support Practice Change in Community Oncology. J Clin Oncol. 2015 Aug 20;33(24):2705-11. doi: 10.1200/JCO.2014.60.6210. Epub 2015 Jul 20. PMID 26195715
- [Background] Minasian LM, Carpenter WR, Weiner BJ, Anderson DE, McCaskill-Stevens W, Nelson S, Whitman C, Kelaghan J, O'Mara AM, Kaluzny AD. Translating research into evidence-based practice: the National Cancer Institute Community Clinical Oncology Program. Cancer. 2010 Oct 1;116(19):4440-9. doi: 10.1002/cncr.25248. PMID 20572032
- [Background] Fiore M, Jaen C, Baker T, Bailey W, Benowitz N, Curry S. Treating Tobacco Use and Dependence: 2008 Update - TreatingTobaccoUseandDependence-2008Update.pdf. http://www.aafp.org/dam/AAFP/documents/patient_care/clinical_recommendations/TreatingTobaccoUseandDependence-2008Update.pdf. Published 2008. Accessed January 11, 2017.
- [Background] Spangler JG, Song EY, Pockey JR, Sutfin EL, Helme DW, Jones C, Foley KL. Predictors of Clinician Tobacco Intervention Counseling in Six North Carolina Free Clinics. Tob Use Insights. 2012 Jul 10;20125:11-16. doi: 10.4137/TUI.S9350. PMID 23843713
- [Background] McNamara RS, Y Song E, Reboussin BA, Spangler J, Pockey JR, Kimes C, Foley KL, Sutfin EL. Motivational interviewing intervention with college student tobacco users: providers' beliefs and behaviors. J Am Coll Health. 2015;63(4):286-90. doi: 10.1080/07448481.2014.1003376. PMID 25580630
- [Background] Lewis JA, Petty WJ, Tooze JA, Miller DP, Chiles C, Miller AA, Bellinger C, Weaver KE. Low-Dose CT Lung Cancer Screening Practices and Attitudes among Primary Care Providers at an Academic Medical Center. Cancer Epidemiol Biomarkers Prev. 2015 Apr;24(4):664-70. doi: 10.1158/1055-9965.EPI-14-1241. Epub 2015 Jan 22. PMID 25613118
- [Background] Foley KL, Farmer DF, Petronis VM, Smith RG, McGraw S, Smith K, Carver CS, Avis N. A qualitative exploration of the cancer experience among long-term survivors: comparisons by cancer type, ethnicity, gender, and age. Psychooncology. 2006 Mar;15(3):248-58. doi: 10.1002/pon.942. PMID 15940742
- [Background] Foley KL, Crandall SJ, George G, Roman M, Spangler JG. Reliability of a Smoking Cessation Risk Factor Interview Scale (SCRFIS) for use with standardized patient instructors. J Cancer Educ. 2003 Fall;18(3):134-41. doi: 10.1207/S15430154JCE1803_06. PMID 14582483
- [Background] Spangler JG, George G, Foley KL, Crandall SJ. Tobacco intervention training: current efforts and gaps in US medical schools. JAMA. 2002 Sep 4;288(9):1102-9. doi: 10.1001/jama.288.9.1102. PMID 12204079
- [Background] Foley KL, Sutfin EL. Availability of tobacco cessation services in free clinics. N C Med J. 2008 Jul-Aug;69(4):270-4. PMID 18828315
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] SRNT Subcommittee on Biochemical Verification. Biochemical verification of tobacco use and cessation. Nicotine Tob Res. 2002 May;4(2):149-59. doi: 10.1080/14622200210123581. No abstract available. PMID 12028847
- [Background] Holt DT, Armenakis AA, Feild HS, Harris SG. Readiness for Organizational Change: The Systematic Development of a Scale. J Appl Behav Sci. 2007;43(2):232-255. doi:10.1177/0021886306295295.
- [Background] Bradley EH, Curry LA, Ramanadhan S, Rowe L, Nembhard IM, Krumholz HM. Research in action: using positive deviance to improve quality of health care. Implement Sci. 2009 May 8;4:25. doi: 10.1186/1748-5908-4-25. PMID 19426507
- [Background] Greenhalgh T, Robert G, Macfarlane F, Bate P, Kyriakidou O. Diffusion of innovations in service organizations: systematic review and recommendations. Milbank Q. 2004;82(4):581-629. doi: 10.1111/j.0887-378X.2004.00325.x. PMID 15595944
- [Background] Greenhalgh T, Robert G, Macfarlane F, Bate P, Kyriakidou O, Peacock R. Storylines of research in diffusion of innovation: a meta-narrative approach to systematic review. Soc Sci Med. 2005 Jul;61(2):417-30. doi: 10.1016/j.socscimed.2004.12.001. Epub 2005 Jan 26. PMID 15893056
- [Background] Kowalski K, Casper C. The coaching process: an effective tool for professional development. Nurs Adm Q. 2007 Apr-Jun;31(2):171-9. doi: 10.1097/01.NAQ.0000264867.73873.1a. PMID 17413512
- [Background] Papadakis S, Pipe AL, Reid RD, Tulloch H, Mullen KA, Assi R, Cole AG, Wells G. Effectiveness of performance coaching for enhancing rates of smoking cessation treatment delivery by primary care providers: Study protocol for a cluster randomized controlled trial. Contemp Clin Trials. 2015 Nov;45(Pt B):184-190. doi: 10.1016/j.cct.2015.08.013. Epub 2015 Sep 5. PMID 26348788
- [Background] Glasgow RE, Green LW, Taylor MV, Stange KC. An evidence integration triangle for aligning science with policy and practice. Am J Prev Med. 2012 Jun;42(6):646-54. doi: 10.1016/j.amepre.2012.02.016. PMID 22608384
- [Background] Newhouse R, Bobay K, Dykes PC, Stevens KR, Titler M. Methodology issues in implementation science. Med Care. 2013 Apr;51(4 Suppl 2):S32-40. doi: 10.1097/MLR.0b013e31827feeca. PMID 23502915
- [Background] Etter JF, Neidhart E, Bertrand S, Malafosse A, Bertrand D. Collecting saliva by mail for genetic and cotinine analyses in participants recruited through the Internet. Eur J Epidemiol. 2005;20(10):833-8. doi: 10.1007/s10654-005-2148-7. PMID 16283473
- [Background] Strecher VJ, McClure J, Alexander G, Chakraborty B, Nair V, Konkel J, Greene S, Couper M, Carlier C, Wiese C, Little R, Pomerleau C, Pomerleau O. The role of engagement in a tailored web-based smoking cessation program: randomized controlled trial. J Med Internet Res. 2008 Nov 4;10(5):e36. doi: 10.2196/jmir.1002. PMID 18984557
- [Background] Bock BC, Papandonatos GD, de Dios MA, Abrams DB, Azam MM, Fagan M, Sweeney PJ, Stein MD, Niaura R. Tobacco cessation among low-income smokers: motivational enhancement and nicotine patch treatment. Nicotine Tob Res. 2014 Apr;16(4):413-22. doi: 10.1093/ntr/ntt166. Epub 2013 Oct 30. PMID 24174612
- [Background] Omar RZ, Thompson SG. Analysis of a cluster randomized trial with binary outcome data using a multi-level model. Stat Med. 2000 Oct 15;19(19):2675-88. doi: 10.1002/1097-0258(20001015)19:193.0.co;2-a. PMID 10986541
- [Background] Schauer GL, Malarcher AM, Asman KJ. Trends in the Average Age of Quitting Among U.S. Adult Cigarette Smokers. Am J Prev Med. 2015 Dec;49(6):939-44. doi: 10.1016/j.amepre.2015.06.028. Epub 2015 Sep 9. PMID 26362404
- [Background] D'Agostino R, Karter A, Lang W, Walkup M, Morgan T. Examining the impact of missing data on propensity score estimation in determining the effectiveness of self-monitoring of blood glucose (SMBG). Health Serv Outcomes Res Methodol. 2001;2:291-315.
- [Background] D'Agostino RB, Rubin DB. Estimating and Using Propensity Scores with Partially Missing Data. J Am Stat Assoc. 2000;95(451):749-759. doi:10.2307/2669455.
- [Background] D'Agostino RB Jr, D'Agostino RB Sr. Estimating treatment effects using observational data. JAMA. 2007 Jan 17;297(3):314-6. doi: 10.1001/jama.297.3.314. No abstract available. PMID 17227985
- [Derived] Foley KL, Dressler EV, Weaver KE, Sutfin EL, Miller DP Jr, Bellinger C, Kittel C, Stone RJ, Petty WJ, Land SR, Spangler JG, Lesser GJ, Chiles C; Optimizing Lung Screening Trial Writing Team. The Optimizing Lung Screening Trial (WF-20817CD): Multicenter Randomized Effectiveness Implementation Trial to Increase Tobacco Use Cessation for Individuals Undergoing Lung Screening. Chest. 2023 Aug;164(2):531-543. doi: 10.1016/j.chest.2023.03.013. Epub 2023 Mar 15. PMID 36931460
- See also: Medicare Coverage Database - Centers for Medicare & Medicaid Services — http://www.cms.gov/medicare-coverage-database/overview-and-quick-search.aspx?FriendlyError=InvalidNCAID
- See also: Bradley EH, Pallas S, Bashyal C, Berman P, Curry L. Developing Strategies for Improving Health Care Delivery : Guide to Concepts, Determinants, Measurement, and Intervention Design. June 2010. — http://openknowledge.worldbank.org/handle/10986/13610
- See also: Johnson. HR at MIT | Learning & Development | What is Coaching? — http://hr.mit.edu/learning-topics/leading/articles/what-is-coaching

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-six radiology facilities in twenty states were selected to participate. Clinics were matched based on lung screening volume and racial/ethnic diversity, and then assigned to the intervention or usual care group. Radiology facilities in the intervention arm participated in multi-faceted implementation strategies targeting the radiology facility and its clinical team. Each clinic was asked to recruit 50 participants.
Pre-assignment Details: Goal was 1100 and there were 6 participants later found to be ineligible due to mis-specified eligibility criteria which is why we have 1094 total.
Groups:
- Intervention: Training of Lung Cancer Screening Personnel on implementation of the US PHS Guidelines for Smoking Cessation and Performance Coaching during Implementation Phase of the Study
  Data collection from Patients: demographics, health status, smoking history, quitting behavior, perceptions of lung cancer risk and worry, impact of screening on tobacco use behavior, and exposure to the intervention. (baseline, <14 days, 3 months, and 6 months)
  Personnel Training and Coaching Calls: Training of Lung Cancer Screening Personnel on implementation of the US PHS Guidelines for Smoking Cessation and Performance Coaching during Implementation Phase of the Study
  Each site will have a coaching team: two members of our research team including an expert in tobacco cessation and an expert in lung cancer screening. Active coaching includes six, 1-1 ½ hour video exchanges among program sites and coaching teams, once every 4-6 weeks over an 8-month implementation phase. One week prior to the call, each site will be prompted with an email to inform the coaching team of any challenges associated with implementation.
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 523 (5 were found ineligible after baseline) | 571 (1 was found ineligible after baseline)
14 Day Follow-up | 483 (32 could not be reached, 1 not interested, 4 too busy to participate, 1 site withdrew, 1 previously consented and removed from study, 1 personal health reasons) | 547 (22 could not be reached, 1 too busy to participate, 1 not interested in participating.)
3 Month Follow-up | 445 (63 could not be reached, 2 refused to answer, 2 expired, 4 not interested in participating, 1 personal health reasons) | 538 (26 could not be reached, 2 expired, and 3 not interested in participating)
Completed | 442 (62 could not be reached, 3 refused to answer, 2 not interested in participating, 1 personal health reason) | 514 (43 could not be reached,2 refused to answer, 2 expired, and 2 not interested in participating)
Not Completed | 81 | 57
Not completed — Lost to Follow-up | 62 | 43
Not completed — Refused to Answer | 5 | 2
Not completed — Death | 2 | 4
Not completed — Not interested in participating | 8 | 6
Not completed — Too busy to participate | 4 | 2

BASELINE CHARACTERISTICS:
Population: 1094 excludes the 6 that were deemed ineligible from the total of 1100 recruited
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 523 | 571 | 1094
Age, Customized [Count of Participants; unit: Participants]
  Age in years: 55-64 | 286 | 333 | 619
  Age in years: 65-74 | 213 | 220 | 433
  Age in years: 75 or older | 24 | 18 | 42
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender, participant reported: Male | 249 | 281 | 530
  Gender, participant reported: Female | 269 | 283 | 552
  Gender, participant reported: Non-Binary | 2 | 3 | 5
  Gender, participant reported: Not Reported | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White, non-Hispanic | 423 | 452 | 875
  Race/Ethnicity: Black, non-Hispanic | 68 | 74 | 142
  Race/Ethnicity: Hispanic, all races | 5 | 23 | 28
  Race/Ethnicity: American Indian, non-Hispanic | 11 | 13 | 24
  Race/Ethnicity: Not Reported | 16 | 9 | 25
Education [Count of Participants; unit: Participants]
  No high school degree, high school degree, or completion of General Education Development (GED) test | 248 | 307 | 555
  Some post high school education or college degree or graduate degree | 272 | 260 | 532
  Not reported | 3 | 4 | 7
Annual Household Income [Count of Participants; unit: Participants]
  Less than $15000 | 94 | 137 | 231
  $15000 - $34999 | 113 | 133 | 246
  $35000 - $64999 | 116 | 116 | 232
  $65000 or higher | 117 | 109 | 226
  Not Reported | 83 | 76 | 159
Marital Status [Count of Participants; unit: Participants]
  Married | 265 | 284 | 549
  Not Currently Married | 254 | 283 | 537
  Not Reported | 4 | 4 | 8
Employment [Count of Participants; unit: Participants]
  Working full- or part-time | 173 | 187 | 360
  Retired | 226 | 226 | 452
  Disabled | 98 | 124 | 222
  Homemaker, Caregiver, Student, or Unemployed | 24 | 31 | 55
  Not Reported | 2 | 3 | 5
Personal Cancer History [Count of Participants; unit: Participants] | 41 | 40 | 81
Family Cancer History [Count of Participants; unit: Participants] | 136 | 165 | 301
Smoke a cigarette within 30 minutes of waking [Count of Participants; unit: Participants] | 372 | 403 | 775
Cigarettes per day [Mean (Standard Deviation); unit: number of cigarettes per day] | 17.3 (10.4) | 17.1 (8.9) | 17.2 (9.6)
Pack Years [Mean (Standard Deviation); unit: pack of cigarettes per day per year] — It is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked.
  pack of cigarettes per day per year | 45.7 (25.7) | 46.5 (24.3) | 46.1 (25.0)
Another smoker in the household [Count of Participants; unit: Participants] | 166 | 158 | 324

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With 7-day Sustained Smoking Abstinence Reported in the Patient Survey
Description: 7-day sustained smoking abstinence will be measured by the question "Have you smoked a cigarette (or other tobacco products), even a puff, in the last 7 days?" in patient survey.
Time Frame: 6 months (after baseline)
Population: Those with completed 6 month surveys.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 442 | 514
percentage of participants | 13.0 [9.7 to 17.4] | 13.5 [10.3 to 17.6]
Statistical Analysis 1: Comparison: Intervention vs Usual Care; A generalized estimating equation marginal model was used in an intent-to-treat analysis to predict the 7-day tobacco use binary outcome. A binomial distribution with logit link was specified with group, time, and the interaction of group by time included as covariates while allowing intercept and time to vary by participants within site with an exchangeable working correlation matrix designation; Test type: Superiority — With 418 analyzable participants across 13 clinics per group, we have 80% power to detect a group difference in primary outcome (7-day abstinence). This assumes control abstinence rate will be 10% versus 20% intervention rate using a 2-sided Z-test for proportions with alpha=0.05 (2-sided). To account for the clustering we used an intra-class correlation value of 0.03. We plan to enroll 1114-1300 patients (or approximately 42-50 per site) to conservatively allow for 25%- 35.5% loss to follow-up; p = 0.865, Mixed Models Analysis; Odds Ratio (OR) = 0.967, 96% CI 2-sided [0.652 to 1.433]

2. Secondary Outcome: Salivary Cotinine Test for Non-Smokers
Description: 7-day Sustained Smoking abstinence will be validated using a salivary cotinine test in non smokers. Abstinence will be determined by percentage of smokers whose tests come back negative for cotinine. Low levels of cotinine less than 15 milligrams per milliliter (mg/mL) would suggest true smoking cessation and levels higher than or equal to 15 mg/mL would suggest they are still smoking.
Time Frame: 6 months (after baseline)
Population: Cotinine was requested only for those that self-reported quitting for at least 7 days at the 6 month survey.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Training of Lung Cancer Screening Personnel on implementation of the United States Public Health Service (US PHS) Guidelines for Smoking Cessation and Performance Coaching during Implementation Phase of the Study
  Data collection from Patients: demographics, health status, smoking history, quitting behavior, perceptions of lung cancer risk and worry, impact of screening on tobacco use behavior, and exposure to the intervention. (baseline, <14 days, 3 months, and 6 months)
  Personnel Training and Coaching Calls: Training of Lung Cancer Screening Personnel on implementation of the US PHS Guidelines for Smoking Cessation and Performance Coaching during Implementation Phase of the Study
  Each site will have a coaching team: two members of our research team including an expert in tobacco cessation and an expert in lung cancer screening. Active coaching includes six, 1-1 ½ hour video exchanges among program sites and coaching teams, once every 4-6 weeks over an 8-month implementation phase. One week prior to the call, each site will be prompted with an email to inform the coaching team of any challenges associated with implementation.
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 51 | 61
Participants
  High: greater than or equal to 15 mg/mL | 13 | 10
  Low: Less than 15 mg/mL | 10 | 20
  Unknown, not tested | 28 | 31

3. Secondary Outcome: Short-term Smoking Abstinence - Patient Survey
Description: Short-tem smoking abstinence will be measured as part of the patient survey as the percentage of patients who report that they have not smoked.
Time Frame: 3 months (after baseline)
Population: Those that had 3 month surveys complete
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 445 | 538
percentage of participants | 6.5 [4.4 to 9.5] | 5.5 [3.8 to 8.0]

4. Secondary Outcome: Total Number of Services Participant Reported Received at 14 Days
Description: Fidelity to the intervention will be measured by a patient survey that asks patients if they received up to 18 cessation services during the screening visit. This is the total each participant reported receiving and can range from 0 to 18, with higher values representing more services.
Time Frame: <= 14 days after baseline
Population: Those that completed 14 day survey
Measure: Least Squares Mean (Standard Deviation); unit: total services reported
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 483 | 547
total services reported | 7.51 (6.33) | 7.86 (6.07)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were not collected as part of this protocol. All-Cause Mortality was not systematically collected or requested, unless a site reported a death when trying to assess the participant at a follow-up visit during the study duration of 6 months and we provide those known cases below.
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/523 | 4/571
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Some sites dropped out early and did not accrue all 50 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT03291587/Prot_SAP_001.pdf
  • Informed Consent Form (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT03291587/ICF_002.pdf